CLINICAL TRIAL: NCT04080518
Title: Hepato-renal Regulation of Water Conservation in Heart Failure Patients With SGLT-2 Inhibitor Treatment
Acronym: DAPA-Shuttle1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2018/2414
Record Dates: First submitted 2019-08-26; First posted 2019-09-06 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: This study will be a 4-week double blind, placebo-controlled, randomized study with 2 treatment arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The assignment of consented patients will occur in a blinded fashion using a randomization scheme generated by a statistician who is not part of the study team and has no contact with the study subject. Once eligibility criteria are met, study participants will be randomly assigned to receive either Dapagliflozin 10mg or matching, identically appearing placebo. Stratified random sampling (by gender) will be performed in order to minimize selection bias. Access to the randomisation code will be controlled and documented. Relevant parties will be blinded to the treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): Dapagliflozin, 10mg, oral dose, once every day
  Interventions: Drug: Dapagliflozin 10 MG [Forxiga]
- Control (Placebo Comparator): Matching placebo for dapagliflozin, oral dose, once every day
  Interventions: Drug: Dapagliflozin 10 MG [Forxiga]

INTERVENTIONS:
Drug: Dapagliflozin 10 MG [Forxiga] — 24 Hour Urine Collection, Sodium (23Na) MRI and Magnetic Resonance (MR) spectroscopy scan, Blood collection for metabolomic and osmolyte analysis
  Other Names: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of Dapagliflozin (FORXIGA) 10mg (n=20) and placebo (n=20) on the renal concentration mechanism, mobilization of Na+ from tissue stores, and mobilization of muscle glycogen and fat, in patients heart failure NYHA classes I and II,with or w/o T2DM in a 4-week double-blind, placebo-controlled, randomized study with 2 treatment arms.

DETAILED DESCRIPTION:
Sodium-glucose co-transporter-2 (SGLT-2) inhibitors are a new class of oral medications used for T2DM, which lower blood glucose levels by increasing renal sodium (Na+) and glucose excretion. However, their applications seem to go beyond glycemic control. Recent studies have shown that treatment with SGLT-2 inhibitors significantly improves cardiovascular outcome, with unprecedented reductions in cardiovascular mortality and heart failure hospitalizations. The underlying mechanism of this surprising effect is unclear.

Our hypothesis is that increased Na+ and glucose excretion induced by SGLT-2 inhibitors predisposes to water loss, to which the body responds by increasing urea production in an effort to prevent dehydration. Urea is accumulated in the renal medulla, where it provides the alternative osmotic driving force for water reabsorption. However, hepatic urea production is an energy-intense process, for which amino acids from skeletal muscle are the ideal fuel because they provide both the nitrogen and the energy needed for urea generation. Alanine is transported from muscle to the liver, where it serves as a substrate for new pyruvate generation, which can then be used for the urea cycle, glucose production or ketone body generation. In the same time, as increasing amounts of alanine are shuttled to the liver, muscle will deplete its glucose reservoirs and reprioritize fuel utilization in favour of fatty acids.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of heart failure NYHA stage I or II - as shown by their medical records
2. Stable anti-hypertensive treatment (>4 weeks)
3. Male and female patients older than 21 years
4. Willingness to participate and ability to provide informed consent
5. Willingness to use effective birth control if of childbearing potential. Any kind of contraception method will be allowed for the period of the study

Exclusion Criteria:

1. Patients with congestive heart failure NYHA stages I (LVEF >40%) without type 2 diabetes mellitus.
2. Patients with congestive heart failure NYHA stages III and IV
3. Prior serious hypersensitivity reaction to Dapagliflozin (Forxiga®)
4. Treatment with any SGLT-2 inhibitor or combined SGLT-1 and 2 inhibitors within 1 week prior to Visit 1 or during screening period until Visit 1
5. Pregnant and breast-feeding women
6. Diagnosis of type 1 diabetes mellitus
7. Patients with type 2 diabetes mellitus with HbA1C > 10.5% from most recent medical records or antidiabetic therapies other than metformin, sulfonylureas or gliptins at screening.
8. Patients with type 2 diabetes mellitus whose antidiabetic treatment (metformin and/or sulfonylureas and/or gliptins) has been changed or unstable within 6 weeks prior to Visit 1
9. . Unstable or rapidly progressing renal disease
10. Chronic cystitis and recurrent urinary tract infections
11. Impaired renal function with eGFR<45 ml/min/1.73m2 or proteinuria > 0.5 g/24h
12. Severe hepatic impairment (Child-Pugh class C)
13. Any major cardiovascular event/vascular disease within 3 months prior to enrolment, as assessed by the investigator
14. Severe edema (as judged by the investigator)
15. Active cancer, history of bladder cancer
16. HIV infection
17. Patients who have received an organ or bone marrow transplant
18. Patients who have had major surgery in the past 3 months
19. Patients who have severe comorbid conditions likely to compromise survival or study participation
20. Patients who exhibit noticeable anxiety and/or claustrophobia or who exhibit severe vertigo when they are moved into the MRI scanner
21. Patients with exclusion criteria for the MRI, such as:

    1. implanted devices (surgical clips, heart pacemakers or defibrillators, cochlear implants)
    2. iron-based tattoos
    3. any other pieces of metal or devices that are not MR-Safe anywhere in the body
22. Unwillingness or other inability to cooperate

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate that SGLT-2 inhibition induces urea-dominated renal water conservation within the renal concentration mechanism. ( Change from baseline in urinary osmolyte concentration | Baseline, Day 3, and Day 28.
  Change from baseline in urinary osmolyte concentration
  1. Change from baseline in Na+
  2. Change from baseline in urea concentration

SECONDARY OUTCOMES:
To demonstrate that SGLT-2 inhibition increases plasma co-peptin levels in an effort to prevent dehydration | Baseline, Day 3 and Day 28
  The investigators will study the changes in plasma co-peptin levels shortly after SGLT-2 inhibitor treatment initiation.
Analysis of skin and muscle Na+ content | Baseline, Day 3, and Day 28.
  The investigators will compare the changes in skin and muscle Na+ content shortly after SGLT-2 inhibitor treatment initiation. Tissue Na+ content will be measured non-invasively with 23NaMRI, using a Siemens 3T MRI scanner system.
Analysis of glycogen and fat content in skeletal muscle and liver | Baseline, Day 3 and Day 28
  The investigators will compare changes from baseline in muscle and liver lipid content (measured with 1HMRS) and assess glycogen content by metabolomic analysis in patients treated with dapagliflozin versus those receiving placebo

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marton A, Saffari SE, Rauh M, Sun RN, Nagel AM, Linz P, Lim TT, Takase-Minegishi K, Pajarillaga A, Saw S, Morisawa N, Yam WK, Minegishi S, Totman JJ, Teo S, Teo LLY, Ng CT, Kitada K, Wild J, Kovalik JP, Luft FC, Greasley PJ, Chin CWL, Sim DKL, Titze J. Water Conservation Overrides Osmotic Diuresis During SGLT2 Inhibition in Patients With Heart Failure. J Am Coll Cardiol. 2024 Apr 16;83(15):1386-1398. doi: 10.1016/j.jacc.2024.02.020. PMID 38599715